CLINICAL TRIAL: NCT03368742
Title: A Randomized, Controlled, Open-label, Single-ascending Dose, Phase I/II Study to Investigate the Safety and Tolerability, and Efficacy of Intravenous SGT-001 in Male Adolescents and Children With Duchenne Muscular Dystrophy
Brief Title: Microdystrophin Gene Transfer Study in Adolescents and Children With DMD
Acronym: IGNITE DMD
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Solid Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GX1001
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SGT-001 - Dose Level 1 (Experimental): Single IV infusion of SGT-001 at starting dose
  Interventions: Genetic: SGT-001
- SGT-001 - Dose Level 2 (Experimental): Single IV infusion of SGT-001 at next ascending dose
  Interventions: Genetic: SGT-001
- Untreated Control (No Intervention): Untreated control group. After 1 year, treatment-eligible control participants will receive SGT-001 at the selected dose.

INTERVENTIONS:
Genetic: SGT-001 — AAV9 vector containing muscle-specific promoter and microdystrophin construct
  Arms: SGT-001 - Dose Level 1; SGT-001 - Dose Level 2

SUMMARY:
This is a controlled, open-label, single-ascending dose study to evaluate the safety and tolerability of SGT-001 in adolescents and children with Duchenne muscular dystrophy (DMD). Participants will receive a single intravenous (IV) infusion of SGT-001 and will be followed for approximately 5 years.

The protocol was amended to drop the control arm after 4 participants were dosed.

ELIGIBILITY:
Inclusion Criteria:

* Established clinical diagnosis of DMD and documented dystrophin gene mutation predictive of DMD phenotype
* Confirmed absence of dystrophin as determined by muscle biopsy (ambulatory participants)
* Anti-AAV9 antibodies below protocol-specified thresholds
* Stable cardiac and pulmonary function
* Adolescents: non-ambulatory by protocol-specified criteria
* Children: ambulatory by protocol-specified criteria
* Stable daily dose (or equivalent) of oral corticosteroids ≥ 12 weeks

Exclusion Criteria:

* Prior or ongoing medical condition or physical examination, ECG or laboratory findings that could adversely affect participant safety, compromise completion of treatment and follow-up, or impair assessment of study results
* Abnormal liver function
* Abnormal renal function
* Clinically significant coagulation abnormalities
* Impaired cardiovascular function based on cardiac MRI or ECHO
* Impaired respiratory function based on FVC % predicted or need for daytime ventilatory support
* Significant spinal deformity or presence of spinal rods
* Body mass index ≥ 95th percentile for age
* Exposure to another investigational drug within 3 months or 5 half-lives prior to screening
* Exposure to drugs affecting dystrophin or utrophin expression within 6 months prior to screening

Additional inclusion/exclusion criteria may apply.

Ages: 4 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 5 years

SECONDARY OUTCOMES:
Number of Participants with Clinically Significant Abnormalities in Laboratory Parameters | Up to 5 years
Number of Participants with Clinically Significant Abnormalities in Vital Signs | Up to 5 years
Number of Participants with Clinically Significant Abnormalities in Physical Examinations | Up to 5 years
Number of Participants with Clinically Significant Abnormalities in Electrocardiogram (ECG) | Up to 5 years
Change from Baseline in Microdystrophin Protein Levels in Muscle Biopsies Using Western Blot (WB) | Baseline, 12 months
Change from Baseline in Microdystrophin Protein Levels in Muscle Biopsies Using Immunofluorescence (IF) | Baseline, 12 months
Change from Baseline in North Star Ambulatory Assessment (NSAA) score in Ambulatory Participants | Baseline, 12 months
Change from Baseline in 6-minute walk test (6MWT) Distance in Ambulatory Participants | Baseline, 12 months
Change from Baseline in Total Upper Limb Function, as Measured by the Total Performance of the Upper Limb (PUL) Functional Scale Score | Baseline, 12 months
Change from Baseline in Respiratory Function, as Measured by Forced Vital Capacity (FVC) % Predicted, Forced Expiratory Volume in 1 second (FEV1) % Predicted, and Peak Expiratory Flow (PEF) % Predicted | Baseline, 12 months
Change from Baseline in Ejection Fraction, As Measured by Echocardiography | Baseline,12 months
Change from Baseline in Left Ventricular End Systolic Volume, As Measured by Echocardiography | Baseline,12 months
Change from Baseline in Myocardial Peak Circumferential Strain (Ecc), As Measured by Echocardiography | Baseline,12 months
Change from Baseline in Quality of Life as Measured by the Paediatric Quality of Life Inventory (PedsQL) Duchenne muscular dystrophy (DMD) module and self-reported outcome measures as measured by the PODCI DMD module | Baseline, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Solid Bio Clinical Trials, Study Director — Solid Biosciences
Locations (2):
- United States (2):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boehler JF, Brown KJ, Ricotti V, Morris CA. N-terminal titin fragment: a non-invasive, pharmacodynamic biomarker for microdystrophin efficacy. Skelet Muscle. 2024 Jan 16;14(1):2. doi: 10.1186/s13395-023-00334-y. PMID 38229112